CLINICAL TRIAL: NCT04356079
Title: Familial and Environmental Factors Behind Migraine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Mohamed Aly Tohamy, Ass. Prof., Assiut University
Other Study IDs: FEFM
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraine patients
  Interventions: Diagnostic Test: International Headache Society Test
- Control
  Interventions: Diagnostic Test: International Headache Society Test

INTERVENTIONS:
Diagnostic Test: International Headache Society Test — Thorough History of Patients and families
  Other Names: Family Pedigree Chart

SUMMARY:
Migraine is a chronic neurological disease characterized by recurrent moderate to severe headaches often in association with a number of autonomic nervous system symptoms. Migraines are believed to be due to a mixture of environmental and genetic factors. About two-thirds of cases run in families. Changing hormone levels may also play a role, as migraines affect slightly more boys than girls before puberty, but about two to three times more women than men after puberty. The risk of migraines usually decreases during pregnancy. The exact mechanisms of migraine are not known. It is, however, believed to be a neurovascular disorder. The primary theory is related to increased excitability of the cerebral cortex and abnormal control of pain neurons in the trigeminal nucleus of the brainstem.

DETAILED DESCRIPTION:
Environmental influences play a role, but family studies suggest that defective genes may be primarily involved in disease causation. The mode of transmission of typical migraine in families is still unclear, but it is widely believed to be multifactorial although a role for a major susceptibility gene cannot be excluded. Aim of study: we aim to study the familial risk for developed migraine and its relation to EEG changes.

ELIGIBILITY:
Inclusion Criteria:

* Fullfilled Migraine chriteria

Exclusion Criteria:

* Genereal Neurologic Disease

Ages: 15 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Patients suffering from Headache between 15 and 45 years old
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of risk factors for migraine | 6 months
  Familial History

IPD SHARING:
Plan to Share IPD: Undecided